CLINICAL TRIAL: NCT03340311
Title: Evaluating the Feasibility of Using M-Health to Improve Serum Glucose Logs of Women With Gestational Diabetes
Brief Title: Evaluating the Feasibility of Using M-Health to Improve Serum Glucose Logs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leslie Balcazar De Martinez (Other)
Responsible Party: Sponsor-Investigator, Leslie Balcazar De Martinez, Doctorate of Nursing Practice Student, University of Virginia
Organization: University of Virginia (Other)
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20100
Record Dates: First submitted 2017-10-20; First posted 2017-11-13 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Gestational Diabetes Mellitus
Keywords: M-Health, GDM, Bluetooth, SMBG
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pre-Post (Other): (Phase one): Each participant will receive usual care (four weeks). Four weeks of glucose logs will be collected at patient's provider visits and completeness recorded.
  (Phase two): Each participant will receive a BG5 wireless glucose meter with supplies enough for four weeks. Each participant will download the iGluco application to their smartphone. Education will be given on the monitor and iGluco application use. Four weeks of glucose logs will be collected at patient's provider visits and completeness recorded.
  At the conclusion of phase 2, the participants will be asked to complete a satisfaction survey about the care received and their preference of monitors.
  Interventions: Device: iHealth Wireless Smart Gluco- Monitoring System (BG5)

INTERVENTIONS:
Device: iHealth Wireless Smart Gluco- Monitoring System (BG5) — Over the course of 8 weeks, participants collected serum glucose logs (SGL) for 4 weeks using usual care followed by SGL's log for 4 weeks using Bluetooth-enabled glucometers and the iGluco application.

SUMMARY:
Gestational diabetes mellitus (GDM) can cause adverse outcomes for the mother and fetus due to hyperglycemia. The purpose of this study is to evaluate the feasibility of improving pregnant women's glucose logs using a Bluetooth enabled glucose monitor and associated mobile health application and to assess their satisfaction with using mobile health technology.

DETAILED DESCRIPTION:
Study Question: Does use of a Bluetooth enabled serum glucose monitor in conjunction with a mobile health application improve pregnant women's glucose log completion? This pilot study proposes that the use of Bluetooth glucometers and mobile health applications will be feasible and well accepted by the target population.

Methods: This project utilizes a quasi-experimental pre-post design with up to 25 participants. Over the course of eight weeks, participants will collect serum glucose logs (SGL) for four weeks using usual care followed by SGLs for four weeks using Bluetooth-enabled glucometers and the iGluco application. Measures will include a demographic sheet and completed SGL. Descriptive statistics of the appropriate level will be used to summarize the data collected. Glucose log completeness will be calculated using the total number of entries required for the period between visits divided by the number of actual entries. For example, if the participant has had 14 days between appointments, 56 entries would be expected, if the patient only records 40 results the completeness score would be 0.71. Raw data will be reported in the final manuscript under results. The data anticipated from this study include the number of women who consented to participate, average education level, primary languages, age range with mean age, the number of women on medication or diet only control, average completion score for usual care phase, and average completion score for the intervention phase. Data will also be generated and reported for the number of patients that did not bring their logs but brought their smartphones or glucometer for transcription and the number of patients that dropped out of the study before completion of eight weeks of glucose logs, and a mean satisfaction score calculated. Eligibility for this study includes women who are at least 18 years old, competent for consent, have gestational diabetes, speak English, have ownership of a smartphone capable of running the mobile health application and are willing to download the application.

Implications: This study has the potential to demonstrate the feasibility of improved Self-management of GDM and provide the groundwork for future studies. The use of Bluetooth enabled glucose monitors with mobile health applications to aid in efficient and complete SMBG management may translate to a decrease in adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

At least 18 years old

* Willing and able to give informed consent
* Diagnosis of gestational diabetes
* Speak English and/or Spanish
* Have ownership of a smartphone capable of running the mobile health application
* Willing to download the iGluco mobile phone application

Exclusion Criteria:

* Have knowledge that their delivery will occur prior to completion of the required eight weeks of glucose logs
* Possess a Bluetooth enabled glucometer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Glucose log completeness | 8 weeks
  Glucose log completeness will be calculated using the total number of entries required for the period between visits divided by the number of actual entries. For example, if the participant has had 14 days between appointments, 56 entries would be expected, if the patient only records 40 results the completeness score would be 0.71.

SECONDARY OUTCOMES:
Patient satisfaction | 1 day at the end of the study.
  Adapted from the PSQ-18 with a question added to determine patients device preference.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Drake, RN, Ph.D, Study Chair — University of Virginia
Locations (1):
- University of Virginia Maternal Fetal Medicine Clinic, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No